CLINICAL TRIAL: NCT03044171
Title: Effect of Sodium Fluoride at 1.1%, Associated or Not With the Low-level Light Therapy in the Prevention of Post-bleaching Sensitivity: a Randomized, Double-blind, Controlled Trial
Brief Title: Evaluation of the Effect of Fluoride and Laser Application on the Prevention of Sensitivity in Bleached Teeth
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Universidade Federal do Para (Other)
Responsible Party: Principal Investigator, Cecy Martins Silva, Associate Professor, Universidade Federal do Para
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: UFPara-001
Record Dates: First submitted 2017-01-30; First posted 2017-02-06 (Estimated); Last update posted 2017-03-17 (Actual); Status verified 2017-03

CONDITIONS: Dentin Sensitivity
MeSH Terms: conditions — Dentin Sensitivity | interventions — Low-Level Light Therapy; Sodium Fluoride; Hydrogen Peroxide

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- G-FLUOR+LASER (Experimental): The corresponding hemiarcade received the application of Low Level Laser Therapy as a desensitizing treatment prior to in-office dental bleaching, followed by the application of 1.1% sodium fluoride after dental bleaching.
  Interventions: Device: Low Level Laser Therapy; Drug: 1.1% Sodium Fluoride; Drug: In-office dental bleaching
- G-FLUOR (Experimental): The correspondent hemiarcade received only the positioning of the inactive laser tip (placebo), prior to in-office dental bleaching, followed by the application of 1.1% sodium fluoride as a desensitizing treatment after dental bleaching
  Interventions: Drug: 1.1% Sodium Fluoride; Drug: In-office dental bleaching

INTERVENTIONS:
Device: Low Level Laser Therapy — Laser therapy: it was used the infrared spectrum with wavelength of 808 nm in its active environment AsGaAl, in two points: cervical and central-medial region of the incisors, canines and premolars.
  Other Names: LLLT
  Arms: G-FLUOR+LASER
Drug: 1.1% Sodium Fluoride — Fluoride therapy: 1.1% sodium fluoride 5000 ppm was applied for 5 minutes on the vestibular surface of all pre-bleached dental elements.
  Other Names: Fluoride therapy
Drug: In-office dental bleaching — Both groups received the in-office bleaching treatment. Three 15-minute applications of the 35% hydrogen peroxide gel were performed, totaling 45 minutes in each of the 4 sessions, with a 7-day interval.
  Other Names: 35% hydrogen peroxide

SUMMARY:
To investigate the effects of desensitizing agents on the dental bleaching process, testing the hypothesis that they may prevent dental sensitivity.

DETAILED DESCRIPTION:
The objective of this double blind, randomized and controlled clinical study, was to evaluate the efficacy of 1.1% sodium fluoride associated with LLLT (Low Level Laser Therapy) on teeth that were exposed to 35% hydrogen peroxide during 4 weeks of bleaching treatment. Methods: 25 volunteers were evaluated through the split-mouth model, where the hemiarcates were ranzomized and later allocated in one of the experimental groups: G-FLUOR+LASER - constitutes the group treated with LLLT + 1.1% sodium fluoride; and G-FLUOR - constitutes the group treated with placebo + 1.1% sodium fluoride .

ELIGIBILITY:
Inclusion Criteria:

* Absence of active carious lesions;
* Good oral hygiene;
* Do not present hypersensitivity;
* Do not smoke;
* Not being pregnant.

Exclusion Criteria:

* Presence of periodontal disease;
* Presence of cracks or fractures;
* Presence of restorations and prostheses;
* Presence of gastroesophageal dysfunction;
* Patients with severe internal dental dimming.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2017-01-23 (Actual); Study Completion 2017-02-23 (Actual)

PRIMARY OUTCOMES:
Stimulated pain intensity measure (P5) | 4 weeks
  Self reported stimulated pain intensity assessed weekly, by modified visual scale, at baseline, after first, second, third and fourth in-office bleaching application. Each item is scored 0-3 (0 = no pain; 3 = pain as bad as can be).

SECONDARY OUTCOMES:
Non-stimulated pain intensity measure, (P28) | 28 days
  Self reported non-stimulated pain intensity, assessed daily, by modified visual scale. Each item is scored 0-3 (0 = no pain; 3 = pain as bad as can be).
Recurrence of stimulated pain | 2 months
  Return of stimulated pain after one month of the last intervention. Item is scored 0-3 (0 = no pain; 3 = pain as bad as can be).

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reis A, Dalanhol AP, Cunha TS, Kossatz S, Loguercio AD. Assessment of tooth sensitivity using a desensitizer before light-activated bleaching. Oper Dent. 2011 Jan-Feb;36(1):12-7. doi: 10.2341/10-148-CR. Epub 2011 Mar 24. PMID 21488723
- [Result] Moosavi H, Arjmand N, Ahrari F, Zakeri M, Maleknejad F. Effect of low-level laser therapy on tooth sensitivity induced by in-office bleaching. Lasers Med Sci. 2016 May;31(4):713-9. doi: 10.1007/s10103-016-1913-z. Epub 2016 Mar 10. PMID 26964798
- Available data/document: Study Protocol: 57655916.3.0000.0018 — http://aplicacao.saude.gov.br/plataformabrasil/visao/pesquisador/gerirPesquisa/gerirPesquisaAgrupador.jsf